CLINICAL TRIAL: NCT05751564
Title: Enabling Advanced Medical Therapy in the Americas: A Pilot Study to Validate a "Ready-to-use" Intra-articular Formulation of Mesenchymal Stromal Cells, Aiming Toward an Effective and Scalable Treatment for Symptomatic Knee Osteoarthritis
Brief Title: "Ready-to-use" Intra-articular Formulation of Mesenchymal Stromal Cells
Acronym: PANLAR-II
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad de los Andes, Chile (Other)
Collaborators: Liga Panamericana de Asociaciones de Reumatologia (PANLAR) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PANLAR-II
Record Dates: First submitted 2023-02-09; First posted 2023-03-02 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-01

CONDITIONS: Osteo Arthritis Knee
Keywords: Osteoarthritis; Degenerative joint disease; Cell therapy; Advanced Medicinal Therapy Product; Mesenchymal Stromal Cell; Mesenchymal Stem Cell; Cryopreserved cell therapy
MeSH Terms: conditions — Osteoarthritis; Joint Diseases | interventions — Pharmaceutical Preparations

STUDY DESIGN:
Intervention Model Description: Prospective Double blind Randomized Controlled Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, providers, investigators and outcome assessments will be blind to randomization except in need to open code for security reasons
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "Ready to inject" MSC product (Experimental): Cryopreserved "ready to inject" Umbilical Cord (UC) derived MSC
  Interventions: Biological: "Ready to inject" Umbilical cord-derived Mesenchymal Stromal Cell (MSC) product
- Resuspended MSC product (Active Comparator): Umbilical Cord (UC) derived MSC in suspension media
  Interventions: Biological: Resuspended Umbilical cord-derived Mesenchymal Stromal Cell (MSC) product

INTERVENTIONS:
Biological: "Ready to inject" Umbilical cord-derived Mesenchymal Stromal Cell (MSC) product — Cryopreserved thaw & inject MSC intra-articular therapy
  Other Names: Cryopreserved "Ready to inject" MSC product
  Arms: "Ready to inject" MSC product
Biological: Resuspended Umbilical cord-derived Mesenchymal Stromal Cell (MSC) product — Cryopreserved resuspended MSC intra-articular therapy
  Other Names: Cryopreserved resuspended MSC product
  Arms: Resuspended MSC product

SUMMARY:
The goal of this clinical trial is to compare a newly developed off-the-shelf cryopreserved "ready to inject" Mesenchymal Stem Cell (MSC) product with the usual MSC preparation the investigators have used in knee osteoarthritis (OA) patients. Since usual MSC therapy requires cell manipulation in GMP (Good Manufacturing Practices)-type facilities, this new formulation would enable wider access to Cell therapy and Multicentric clinical trials in areas devoid of expensive facilities and equipment.

DETAILED DESCRIPTION:
This is a double blind randomized controlled trial testing a modified formulation of an allogenic Umbilical cord (UC) derived MSC therapy that the investigators have used in a prior published clinical trial. It has been modified and characterized according to the standards of quality control that are required for the development an off-the-shelf cryopreserved MSCs product.

This so called "ready to inject" MSC preparation will be compared with the usual MSC formulation that requires centrifugation and resuspension in different media, thus requiring access to advanced (GMP-type) facilities.

A total of 60 symptomatic knee OA patients will be randomized (1.1 ratio) to receive one or the other MSC product at baseline and month 6, to be followed blindly for 12 months with baseline and end of study knee MRI imaging.

The primary endpoint of the trial will be the safety according to the occurrence of adverse events (AEs) as coded by the Common Terminology Criteria for Adverse Event classification. The secondary endpoint will be efficacy, as assessed by the following validated clinical outcome measures: Western Ontario and Mc Master Universities Arthritis Index (WOMAC) Spanish validated version, Pain Visual Analog scale (VAS), Quality of life by the Short-form 36 (SF-36) questionnaire, Patient Global Assessment, and the Outcome Measures in Rheumatology Committee (OMERACT)-Osteoarthritis Research Society International (OARSI) Responder Index Criteria. Baseline MRI will be performed mainly to exclude meniscal lesions associated with accelerated knee OA. Final (12 month) MRI will be performed to assess structural change in response to treatment

The completion of this project represents a main technological advance, eventually leading to the scalability and enhanced quality control of a much needed treatment, within reasonable costs and logistics, and in particular, with no need of a GMP facility at the point of care or of clinical testing

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic knee OA defined by grade 1-3 Kellgren-Lawrence radiographic changes in the targeted knee.
* Daily pain at the affected joint for at least 3 months before inclusion

Exclusion Criteria:

* Bilateral symptomatic knee OA (only if the contralateral knee has more severe disease)
* Meniscal rupture.
* Condylar or tibial plateau generalized bone marrow edema on MRI
* Major axial deviation defined by valgus (>10°) or varus (5°) deformity of the involved leg
* Use of oral or intra-articular steroids or hyaluronic acid in the past 6 months
* Ipsilateral hip or ankle pain, local or systemic infection
* Any form of secondary arthritis, previous malignancy, or body mass index ≥30.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-04 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Safety monitoring for Adverse events | 12 months
  Adverse events (AEs) reported for each study group as coded by the Common Terminology Criteria for Adverse Event classification.

SECONDARY OUTCOMES:
WOMAC scale | 12 months
  Western Ontario and Mc Master Universities Arthritis Index (WOMAC) Spanish validated version. Scale ranges from 0-240 with higher scores indicating worsened state
Pain Visual Analog Scale (VAS) | 12 months
  VAS scale for pain, ranging from 0-10 with higher scores indicating worsened state
Quality of Life SF-36 questionnaire | 12 months
  Short-form 36 (SF-36) questionnaire, ranging from 0-100 with higher scores indicating better health status
Responder status | 12 months
  Assessed by the Outcome Measures in Rheumatology Committee (OMERACT)-Osteoarthritis Research Society International (OARSI) Responder Index Criteria. Responder status requires fulfilling at least 50% improvement in pain or function with absolute change of at least 20; or at least 20% improvemente in pain, function or patient´s global assessment, with absolute change of at least 20.

OTHER OUTCOMES:
WORMS SCORE | 12 months
  Baseline and 12 month MRI will be performed to assess structural change in response to treatment as computed by the Whole-Organ Magnetic Resonance Imaging Score (WORMS) of the knee in osteoarthritis. This score ranges 14 imaging features from 0-332 with higher scores indicating worsened state

CONTACTS AND LOCATIONS:
Overall Officials: Fernando E Figueroa, M.D., Principal Investigator — Universidad de Los Andes

IPD SHARING:
Plan to Share IPD: Yes
Sharing upon request after publication of the trial.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: At trial termination and publication.
Access Criteria: Data will be shared with researchers or scholars with no conflict of interest and once we have confirmed the data are not subject to confidentiality due to intellectual property or other issues.

REFERENCES:
- [Background] Matas J, Orrego M, Amenabar D, Infante C, Tapia-Limonchi R, Cadiz MI, Alcayaga-Miranda F, Gonzalez PL, Muse E, Khoury M, Figueroa FE, Espinoza F. Umbilical Cord-Derived Mesenchymal Stromal Cells (MSCs) for Knee Osteoarthritis: Repeated MSC Dosing Is Superior to a Single MSC Dose and to Hyaluronic Acid in a Controlled Randomized Phase I/II Trial. Stem Cells Transl Med. 2019 Mar;8(3):215-224. doi: 10.1002/sctm.18-0053. Epub 2018 Dec 28. PMID 30592390